CLINICAL TRIAL: NCT06524869
Title: Association of Strength and Proprioception Parameters With Qualitative Assessment of Functional Tasks After ACL Reconstruction
Brief Title: Association Between Neuromuscular Parameters and Functional Assessment After ACL Reconstruction
Acronym: KASTLAB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Associate Professor, University Hospital, Caen
Other Study IDs: KASTLAB
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ACL reconstruction group: All sports patients who had a muscle evaluation at 6 to 12 months after ACLR since March 2024
  Interventions: Diagnostic Test: Isokinetic neuromuscular assessment

INTERVENTIONS:
Diagnostic Test: Isokinetic neuromuscular assessment — All sports patients who had a muscle evaluation in addition to functional testing at 6-12 months after ACLR since March 2024

SUMMARY:
The anterior cruciate ligament (ACL) injury is common in athletes aged 18 to 35. ACL reconstruction (ACLR) aims to restore knee stability in the process of returning to sports. Post-surgical rehabilitation focuses on optimizing biomechanical parameters, with neuromuscular and functional tests assessing muscle strength, proprioception, and dynamic stability. Isokinetic allows the measurement of muscle strength symmetry and proprioception, while the single-leg hop and landing tasks assess functional stability and are predictive of sports resumption and injury prevention. Despite progress, concerns remain about neuromuscular factors impacting knee stability, especially during landings, which can increase the risk of secondary ACL injuries.

This study proposes examining knee strength and proprioception using isokinetic dynamometry, alongside biomechanical assessments from functional tests, to explore their relationship to biomechanical features during landings, at 6-to-12 months post-ACL reconstruction. The hypothesis is that better muscle strength and proprioception correlate with improved knee control during landing tasks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, aged 18-40, who have undergone a first ACL reconstruction more than 6 months ago and are being followed in a sports medicine care pathway
* Affiliated with a health insurance plan
* Information form: Non-objection to the use of data for research purposes

Exclusion Criteria:

* Previous ligament surgery of the lower limbs prior to ACL reconstruction
* Complex ligament injury (lateral ligaments, posterior cruciate ligament)
* Recent muscle injuries
* History of injury to the uninjured knee
* Pregnant woman
* Neurological history with residual effects or taking medication that affects balance/coordination
* Inability to perform a muscular assessment
* Postoperative complications (deep vein thrombosis, sepsis, stiffness/arthrofibrosis)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All sports patients included in the sport medicine follow-up protocole with isokinetic muscular assessment at 6-12 months after ACL reconstruction surgery since March 2024 in the sports medicine department (Return To Sport Process)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Passive proprioceptive evaluation | One measurement during the visit at 6 to 12 months after surgery
  Measurement of knee proprioception by the passive repositioning technique (JPS, in degrees) on isokinetic dynamometer.
Strength | One measurement during the visit at 6 to 12 months after surgery
  Measurement of knee extensors and flexors peak strength (in newton.meter, Nm) on isokinetic dynamometer.
Single Hop test | One measurement during the visit at 6 to 12 months after surgery
  Measurement of knee position during landing from a single leg hop task
Single-leg landing task | One measurement during the visit at 6 to 12 months after surgery
  Measurement of knee position during landing from a 30-cm box

SECONDARY OUTCOMES:
Single Hop for Distance | One measurement during the visit at 6 to 12 months after surgery
  The total distance is recorded (in cm)
ACL-RSI questionnaire (Anterior Cruciate Ligament-Return to Sport after Injury) | One measurement during the visit at 6 to 12 months after surgery
  The ACL-RSI measures the patient's understanding of his knee. It comprises 12 questions with a score of 1 to 10 for each
Landing Error Scoring System (LESS) | One measurement during the visit at 6 to 12 months after surgery
  The LESS (Landing Error Scoring System) scale is a 13-item tool used to assess landing technique during a hop task.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Faivre O, Prum G, Hulet C, Drigny J. Improved hamstring strength and knee position sense are associated with enhanced landing mechanics after anterior cruciate ligament reconstruction. J ISAKOS. 2025 Jun;12:100858. doi: 10.1016/j.jisako.2025.100858. Epub 2025 Apr 5. PMID 40194659